CLINICAL TRIAL: NCT07023276
Title: Agility and Movement Quality Among High School Basketball Players Following a Coach-Led Neuromuscular Training Program
Brief Title: Agility and Performance Among High School Basketball Players Following a Coach-Led Neuromuscular Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-1571
Record Dates: First submitted 2025-06-03; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Athletic Performance
Keywords: NMT; neuromuscular training; basketball; movement control; agility; movement mechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromuscular Training Programming (Experimental): Coaches implemented neuromuscular training at the start of all warm-ups for practices and games.
  Interventions: Other: Neuromuscular Training

INTERVENTIONS:
Other: Neuromuscular Training — Coaches implemented neuromuscular training at the start of all warm-ups for practices and games. The neuromuscular training program was developed by sports medicine professionals at the home institution and the National Basketball Association and incorporates established principles of motor learning and performance training and has an added emphasis of being basketball-specific.

SUMMARY:
The purpose of this study is to examine changes in agility and athletic performance of high school basketball players following a coach-led neuromuscular training program. Outcomes were measured at pre- and post-season data collection sessions. Additionally, player attendance and warm-up adherence was self recorded by coaches.

DETAILED DESCRIPTION:
This study recruited high school basketball teams from the greater New York City area. Coaches from the participating teams were trained to implement a neuromuscular training program to their players at the start of a warm-up prior to all practices and games for the duration of their basketball season (10-14 weeks). At pre-season and post-season data collection sessions, players completed agility and movement quality testing. Agility was measured by the Lane Agility Test (LAT) and movement quality testing was measured through completing a series of single leg squats. The single leg squats were recorded and analyzed using a previously scoring criteria (Di Paolo et al. 2024). After videos were analyzed, players were given an overall movement quality score using the scoring criteria.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18 years old
* Active participant on a high school level basketball team with a coach/coaches fluent in English
* Completion of pre- and post-season testing

Exclusion Criteria:

- Individuals who did not complete pre- or post-season testing

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Lane Agility Test (LAT) | Agility was measured at a baseline testing date and then again at the cumulation of the basketball season (duration of 10-14 weeks).
  The lane agility was performed according to previously published methods (Stojanović et al. 2019). The LAT was set up around the basketball court using small cones. Players started at the bottom left corner of the key underneath the basket and sprinted to the cone on the left corner of the free throw line. Players side shuffled to the right, across the free-throw line to the next cone (on the right corner of the free throw line) and then backpedaled towards the third cone at the baseline. Next, the players side-shuffled towards the original cone. Once the player's left foot went past the cone, they re-traced the same route back in the opposite direction. Time was recorded from the moment the player started the course at the bottom left key until the time that the player's entire body backpedaled across the same baseline cone.

SECONDARY OUTCOMES:
Movement Quality | Movement quality was measured at a baseline testing date and then again at the cumulation of the basketball season (duration of 10-14 weeks).
  Players completed a series of six single leg squats on each leg as instructed by sports medicine professionals. All of the squats were recorded on video. For each leg, three of the squats were completed facing towards the camera. The other three squats were completed facing towards the side so that the player's sagittal profile was recorded. The videos were analyzed and annotated with measurements to compute to a single score describing their movement quality as outlined in a previously published scoring criteria (Di Paolo et al. 2024). The overall score ranged from 0 to 8, with a higher score indicating a better performance.
Injury | Duration of the basketball season (expected duration 10-14 weeks).
  Attendance was taken for each player for the duration of the season. Coaches categorized each day of the season as one of the following: "Practice," "Game," or "Off Day." Coaches also indicated if the team completed the neuromuscular training warm-up for the days in which they had practices or games. For each player, coaches took attendance every day and indicated one of the following for practices and games: "Present," "Absent - Excused," "Absent - Unexcused," "Absent - Injury." Injury was defined as the days in which the player was marked "Absent - Injury."

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pearle, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stojanovic E, Aksovic N, Stojiljkovic N, Stankovic R, Scanlan AT, Milanovic Z. Reliability, Usefulness, and Factorial Validity of Change-of-direction Speed Tests in Adolescent Basketball Players. J Strength Cond Res. 2019 Nov;33(11):3162-3173. doi: 10.1519/JSC.0000000000002666. PMID 29927890
- [Background] Di Paolo S, Musa F, d'Orsi GM, Grassi A, Vulpiani MC, Zaffagnini S, Della Villa F. A comprehensive two-dimensional scoring system to assess the single-leg squat task in football players. Knee. 2024 Jun;48:52-62. doi: 10.1016/j.knee.2024.02.016. Epub 2024 Mar 20. PMID 38513322